CLINICAL TRIAL: NCT04691284
Title: Microbiome in Cancer Patients Undergoing High Dose Chemotherapy With Stem Cell Transplantation
Brief Title: Microbiome in Cancer Patients With High Dose Chemotherapy With Stem Cell Transplantation
Acronym: SCTMICROBIOM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Slovakia (Other Government)
Collaborators: Slovak Academy of Sciences (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: PROBIO - SK - 006
Record Dates: First submitted 2020-12-19; First posted 2020-12-31 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Hematologic Neoplasms
Keywords: Cancer; microbiome; high dose chemotherapy; stem cell transplantation; CAR-T cell
MeSH Terms: conditions — Hematologic Neoplasms; Neoplasms | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Observational arm (Experimental): Patients will be asked to provide a sample of blood, urine and stool. This blood will be used for plasma and serum banking for further analysis, including miR and chemokine detection. Stool will be used for microbiome studies - isolation of total DNA/RNA and 16S rRNA gene sequencing for bacterial taxonomic classification. Furthermore, metagenomic sequencing and subsequent taxonomic and functional classification of microbial genes will be used. Moreover, we might be able to characterized potentially clinically relevant features of the microbiome such as antibiotic resistance and microbial virulence factors.
  Interventions: Other: Blood, urine and stool sampling

INTERVENTIONS:
Other: Blood, urine and stool sampling — Sampling of blood and urine for miR and chemokine detection. Sampling of stool for for microbiome studies.

SUMMARY:
Numerous in vitro and animal studies as well as growing number of clinical studies support the important role of microbiome in carcinogenesis and cancer treatment. Detection of changes in patients´ microbiome following hematopoietic cell transplantation/CAR-T cell therapy and correlations with adverse transplant outcomes, mainly infectious complications, acute and chronic GvHD, disease recurrence etc. could serve as predictive markers of immune recovery and treatment response.

DETAILED DESCRIPTION:
Currently, available findings coming mainly from allo-HSCT (hhematopoietic cell transplantation) studies, link particular changes in microbiota with overall survival and post-transplant disorders, especially GvHD. According to limited data, further evaluation of associations between the alterations in microbiome composition and toxicities. Detail investigation of both the microbiome and host immune system may help to find microbiome markers useful for very early identification of patients at risk for major transplant-related complications. This might bring the possibility to modulate the gut microbiota in patient´s specific manner to achieve optimal therapeutic outcome and follow-up, while avoiding severe post-transplant complications.

This is prospective, single center, non-randomized, hypothesis generating study. Patients will be asked to provide a sample of blood, urine and stool. This blood will be used for plasma and serum banking for further analysis, including micro RNA (miR) and chemokine detection. Stool will be used for microbiome studies - isolation of total DNA/RNA and 16S (RNA component of the small subunit of a prokaryotic ribosome) rRNA (ribosomal ribonucleic acid) gene sequencing for bacterial taxonomic classification. Furthermore, metagenomic sequencing and subsequent taxonomic and functional classification of microbial genes will be used including characterization of potentially clinically relevant features of the microbiome such as antibiotic resistance and microbial virulence factors.

ELIGIBILITY:
Inclusion Criteria:

* signed written informed consent
* aged 18 years or older
* patients planned to be treated by high-dose chemotherapy and hematopoietic cell transplantation or by CAR-T cell therapy in National Cancer Institute, Slovakia

Exclusion Criteria:

- patients not-matching inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Microbial changes in stool as measured by 16S rRNA gene sequencing in hematological cancer patients before, at time and after hematopoietic cell transplantation and CAR-T cell therapy | 100 days
  Microbial changes of stool will be assessed before, at time and after hematopoietic cell transplantation and CAR-T cell therapy

SECONDARY OUTCOMES:
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the post-transplant complications in auto and allogeneic transplant settings (GvHD, diarrhea, infectious complications) and in CAR-T cell therapy | 100 days
  To assess microbial changes with toxicity of therapy
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the patients reported outcomes. | 100 days
  To correlate microbial changes with the quality of life, spirituality, cognitive functions
To correlate microbial changes in stool as measured by 16S rRNA gene sequencing with the patients nutrition status | 100 days
  To correlate microbial changes with the patients nutrition.

CONTACTS AND LOCATIONS:
Overall Officials: Luboš Drgoňa, Assoc. Prof., Study Chair — National Cancer Institute, Slovakia; Michal Mego, prof., Study Chair — National Cancer Institute, Slovakia
Locations (1):
- National Cancer Institute, Bratislava, Slovakia, Slovakia

IPD SHARING:
Plan to Share IPD: No